CLINICAL TRIAL: NCT01755546
Title: A Phase 3, Open-label, Long-term Study to Evaluate the Safety, Tolerability, and Analgesic Efficacy of BEMA® Buprenorphine in Subjects With Moderate to Severe Chronic Pain Requiring Continuous Around-the-Clock Opioid Analgesia for an Extended Period of Time
Brief Title: Long-term Open-Label Safety Study to Evaluate EN3409
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: BioDelivery Sciences International (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EN3409-309
Record Dates: First submitted 2012-12-19; First posted 2012-12-24 (Estimated); Results first posted 2018-09-12 (Actual); Last update posted 2018-10-18 (Actual); Status verified 2018-03

CONDITIONS: Low Back Pain; Osteoarthritis; Neuropathic Pain
Keywords: Chronic Pain; CLBP; Chronic Low Back Pain; Back Pain; Osteoarthritis; OA; Neuropathic Pain; Nerve pain; Painful neuropathy
MeSH Terms: conditions — Low Back Pain; Osteoarthritis; Neuralgia; Chronic Pain; Back Pain; Neuropathy, Painful

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- EN3409 (Experimental): Buprenorphine HCI Buccal File at doses ranging from 300-900 mcg twice daily
  Interventions: Drug: EN3409

INTERVENTIONS:
Drug: EN3409 — Open-Label Buprenorphine HCI Buccal Film at doses 300-900 mcg twice daily
  Other Names: Buprenorphine HCI Buccal Film 300-900 mcg twice daily

SUMMARY:
The purpose of the long-terms study is to evaluate the safety, tolerability, and analgesic efficacy of EN3409 in subjects with moderate to severe chronic pain requiring continuous around-the-clock opioid analgesia for an extended period of time.

ELIGIBILITY:
Inclusion Criteria:

* Female subjects who are practicing abstinence or using a medically acceptable form of contraception or have been postmenopausal, biologically sterile, or surgically sterile for more than 1 year
* Male subjects who are practicing abstinence, surgically sterile, or are using a medically acceptable form of contraception
* De Novo subject with a clinical diagnosis of moderate to severe noncancer-related CP (eg, CLBP, OA, neuropathic pain) for ≥ 3 months
* De Novo subject that is treating their CP with a stable daily maintenance dose of ATC opioid analgesic medication equivalent to ≥ 60 mg and ≤ 160 mg Morphine Sulfate Equivalent (MSE) per day for ≥ 4 weeks
* Stable health, as determined by the Principal Investigator
* Subject is willing and able to comply with all protocol required visits and assessments
* Rollover subject who has completed the 12-week Double-blind Treatment Phase in the EN3409-307/308 clinical study

Exclusion Criteria:

* A history or current evidence of any clinically significant disorder or any other condition, which in the opinion of the investigator, would jeopardize the safety of the subject or impact the validity of the study results
* Females who are pregnant, breastfeeding, or plan to become pregnant during the study
* Current cancer-related pain or received chemotherapy within 6 months of screening
* Subjects receiving opioid analgesic medication < 60 mg MSE per day within 28 days of screening
* De novo subjects receiving opioid analgesic medication at doses of > 160 mg MSE per day within 28 days of screening
* Subjects with a history of other chronic painful conditions, other than the index CP condition, which require frequent analgesic medication
* Reflex sympathetic dystrophy or causalgia (complex regional pain syndrome), acute spinal cord compression, cauda equina compression, acute nerve root compression, meningitis, or discitis
* History of allergy or contraindications to any opioid or acetaminophen
* Surgical procedure for relief of pain within 6 months, or nerve/plexus block within 28 days of screening
* Hypokalemia or clinically unstable cardiac disease
* Moderate to severe hepatic impairment
* Moderate to severe renal impairment
* Current or past history of alcohol or substance
* Positive urine toxicology screen for drugs of abuse
* History of abnormalities on physical exam, vital signs, ECG, or lab values

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 304 (Actual)
Dates: Start 2012-12; Primary Completion 2014-10 (Actual); Study Completion 2014-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Finn, PharmD, Study Director — BioDelivary Sciences Internantional, Inc.
Locations (57):
- United States (57):
  - Parkway Medical Center, Birmingham, Alabama
  - Horizon Research Group, Inc, Mobile, Alabama
  - Arizona Research Center, Phoenix, Arizona
  - Global Research, LLC, Anaheim, California
  - Synergy Clinical Research Center of Escondido, Escondido, California
  - RX Clinical Research, Inc., Garden Grove, California
  - Long Beach Center for Clinical Research, Long Beach, California
  - Adam D. Karns, MD, Los Angeles, California
  - Stamford Therapeutics Consortium, Stamford, Connecticut
  - Clinical Research of West Florida, Inc., Clearwater, Florida
  - Century Clinical Research, Inc., Daytona Beach, Florida
  - Avail Clinical Research, LLC, DeLand, Florida
  - Florida Health Center, Fort Lauderdale, Florida
  - Eastern Research, Inc., Hialeah, Florida
  - Southeast Clinical Research, LLC, Jacksonville, Florida
  - Health Awareness, Inc., Jupiter, Florida
  - Research Centers of America, LLC, Oakland Park, Florida
  - Compass Research, LLC, Orlando, Florida
  - Ribo Research LLC DBA Peninsula Research, Ormond Beach, Florida
  - Gold Coast Research, LLC, Plantation, Florida
  - Progressive Medical Research, Port Orange, Florida
  - Clinical Research of West Florida, Inc., Tampa, Florida
  - Palm Beach Research Center, West Palm Beach, Florida
  - National Pain Research Institute, LLC, Winter Park, Florida
  - River Birch Research Alliance, LLC, Blue Ridge, Georgia
  - Drug Studies America, Marietta, Georgia
  - Taylor Research, LLC, Marietta, Georgia
  - In-Quest Medical Research, LLC, Norcross, Georgia
  - Global Scientific Innovations, Evansville, Indiana
  - Integrated Clinical Trials Services, Inc., West Des Moines, Iowa
  - Willis-Knighton Physician Network, Bossier City, Louisiana
  - Clinical Trials Management, LLC, Metairie, Louisiana
  - Best Clinical Trials, LLC, New Orleans, Louisiana
  - River Cities Clinical Research Center, Shreveport, Louisiana
  - New England Center for Clinical Research, Inc., Fall River, Massachusetts
  - Great Lakes Research Group, Inc., Bay City, Michigan
  - Cadillac Clinical Research, Cadillac, Michigan
  - The Center for Clinical Trials, Biloxi, Mississippi
  - Long Island Gastrointestinal Research Group, Great Neck, New York
  - Upstate Clinical Research Associates, Williamsville, New York
  - The Center for Clinical Research, Winston-Salem, North Carolina
  - Plains Medical Clinic, LLC, Fargo, North Dakota
  - Clinical Inquest Center, Ltd, Beavercreek, Ohio
  - New Horizons Clinical Research, Cincinnati, Ohio
  - Prestige Clinical Research, Franklin, Ohio
  - Optimed Research, Ltd., Tiffin, Ohio
  - Brandywine Clinical Research, Downingtown, Pennsylvania
  - Altoona Center for Clinical Research, Duncansville, Pennsylvania
  - Pain Specialists of Charleston, P.A., Charleston, South Carolina
  - Health Concepts, Rapid City, South Dakota
  - FutureSearch Clinical Trials, Austin, Texas
  - KRK Medical Research, Dallas, Texas
  - FutureSearch Trials of Dallas, LP, Dallas, Texas
  - Advanced Clinical Research of Houston, Houston, Texas
  - Innovative Clinical Trials, San Antonio, Texas
  - Highland Clinical Research, Salt Lake City, Utah
  - Clinical Investigations Specialist, Inc., Kenosha, Wisconsin

RESULTS

PARTICIPANT FLOW:
Groups:
- Overall: All subjects combined, Roll Over and De Novo.
Period: Screened and Taper (Rollover and DeNovo)
Arm/Group | Overall
Started | 304
Completed | 294
Not Completed | 10
Not completed — Protocol Violation | 1
Not completed — Withdrawal by Subject | 3
Not completed — Lost to Follow-up | 1
Not completed — Any other reason and screen failures | 5
Period: Titration Phase
Arm/Group | Overall
Started | 294
Completed | 224
Not Completed | 70
Not completed — Adverse Event | 11
Not completed — Lack of Efficacy | 18
Not completed — Protocol Violation | 9
Not completed — Lost to Follow-up | 2
Not completed — Other and Continuing | 22
Not completed — Withdrawal by Subject | 8
Period: Long Term Treatment
Arm/Group | Overall
Started | 224
Completed | 103
Not Completed | 121
Not completed — Adverse Event | 12
Not completed — Lack of Efficacy | 6
Not completed — Protocol Violation | 10
Not completed — Withdrawal by Subject | 35
Not completed — Lost to Follow-up | 17
Not completed — other and ongoing | 41

BASELINE CHARACTERISTICS:
Population: Baseline at start of Long-Term Treatment Phase
Groups:
- Overall: All subjects combined, Roll Over and De-Novo.
Arm/Group | Overall
Number analyzed (Participants) | 224
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 193
  >=65 years | 31
Age, Continuous [Mean (Standard Deviation); unit: Years] | 52 (11.80)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 125
  Male | 99
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 39
  Not Hispanic or Latino | 185
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3
  Asian | 6
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 57
  White | 158
  More than one race | 0
  Unknown or Not Reported | 0
Weight (kg) [Mean (Standard Deviation); unit: kilograms] | 92.2 (21.57)
Height (cm) [Mean (Standard Deviation); unit: centimeters] | 169.5 (10.39)
BMI (kg/m^2) [Mean (Standard Deviation); unit: kg/m^2] | 32.1 (7.20)
NRS Pain Intensity [Mean (Standard Deviation); unit: units on a scale] — The NRS Pain intensity score is a segmented version of a visual analog scale used to measure pain. The scale is from 0 (no pain) to 10. Scores between greater than 0 and 3 are considered mild pain, scores from greater than 3 to 6 are moderate and greater than 6 to 10 are severe. The daily average is calculated and used as baseline.
  units on a scale | 3 (1.30)
Chronic Pain [Count of Participants; unit: Participants]
  Lower Back Pain | 222
  Neuropathic Pain | 1
  Osteoarthritis | 1

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to Week 48 in Daily Average NRS Pain Intensity Score
Description: The NRS Pain intensity score is a segmented version of a visual analog scale used to measure pain. The scale is from 0 (no pain) to 10. Scores between greater than 0 and 3 are considered mild pain, scores from greater than 3 to 6 are moderate and greater than 6 to 10 are severe. The daily average is calculated and the change from baseline at week 48 is presented.
Time Frame: 48 weeks
Population: Efficacy Population
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Overall
Number analyzed (Participants) | 97
units on a scale | 0.2 (1.78)

ADVERSE EVENTS:
Time Frame: 48 Weeks
Arm/Group | Overall
Serious Adverse Events (participants affected / at risk) | 12/224
Other Adverse Events (participants affected / at risk) | 115/224
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Overall (N=224)
Bronchitis (Infections and infestations) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
Urosepsis (Infections and infestations) | 1 (1)
Syncope (Nervous system disorders) | 1 (1)
Status migrainosus (Nervous system disorders) | 1 (1)
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 1 (1)
Renal impairment (Renal and urinary disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Influenza like illness (General disorders) | 1 (1)
Ankle Fracture (Injury, poisoning and procedural complications) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Overall (N=224)
Upper respiratory tract infection (Infections and infestations) | 14 (14)
Bronchitis (Infections and infestations) | 9 (9)
Nasopharyngitis (Infections and infestations) | 7 (7)
Nausea (Gastrointestinal disorders) | 18 (18)
Vomiting (Gastrointestinal disorders) | 11 (11)
Diarrhea (Gastrointestinal disorders) | 10 (10)
Constipation (Gastrointestinal disorders) | 9 (9)
Headache (Nervous system disorders) | 12 (12)
Back pain (Musculoskeletal and connective tissue disorders) | 13 (13)
Fall (Injury, poisoning and procedural complications) | 7 (7)
Depression (Psychiatric disorders) | 8 (8)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No